CLINICAL TRIAL: NCT00646100
Title: Transarterial Chemoembolization Versus Best Support for Unresectable Hepatocellular Carcinoma With Portal Vein Tumor Thrombosis
Brief Title: Transarterial Chemoembolization for Unresectable Hepatocellular Carcinoma With Portal Vein Tumor Thrombosis
Acronym: TACEHCC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Shi Ming, Professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TACE1
Record Dates: First submitted 2008-03-25; First posted 2008-03-28 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; transcatheter arterial chemoembolization; prospective control study; best support care; survival
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TACE (Active Comparator): chemo-lipiodolization with EADM 50mg, Lobaplatin 50mg, and MMC 6mg,plus particleembolization
  Interventions: Procedure: transcatheter arterial chemoembolization
- control (No Intervention): best support care

INTERVENTIONS:
Procedure: transcatheter arterial chemoembolization — chemo-lipiodolization with EADM 50mg, Lobaplatin 50mg, and MMC 6mg,plus particleembolization.
  Other Names: TACE
  Arms: TACE

SUMMARY:
Transcatheter arterial chemoembolization (TACE) had been proved to improve the survivals for middle stage hepatocellular carcinoma (HCC), but for advanced stage HCC its' efficacy had not been proved. The investigators hypothesize that TACE also improve the survivals for advanced stage HCC. Thus, the investigators carried out this prospective control study to find out if the survivals for patients after TACE better than only best support or not.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of HCC was based on the diagnostic criteria for HCC used by the European Association for the Study of the Liver (EASL)
* Tumor size >7 cm with a portal vein invasion, and the tumor was considered to be unresectable
* No previous HCC directed treatment
* Eastern Co-operative Group performance status 0-1
* Liver function: Child's A

Exclusion Criteria:

* Avascular tumor
* Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
* underlying serve cardiac or renal diseases
* Known or suspected allergy to the investigational agent or any agent given in association with this trial
* Diffuse-type HCC
* For patients with main portal vein occlusion, no adequate collateral circulation around the occluded portal vein

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2007-07; Primary Completion 2009-07 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
survival rates | 6, 12 months

SECONDARY OUTCOMES:
quality of life | 6, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: jinqing li, MD, Study Director — cancer canter sun yat-set university
Locations (1):
- Cancer Canter Sun Yat-Sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Bruix J, Sherman M; Practice Guidelines Committee, American Association for the Study of Liver Diseases. Management of hepatocellular carcinoma. Hepatology. 2005 Nov;42(5):1208-36. doi: 10.1002/hep.20933. No abstract available. PMID 16250051